CLINICAL TRIAL: NCT02198365
Title: Comparison of Human Papillomavirus Integrated DNA and Messenger RNA for Detection and Prediction in Progression of Cervical Neoplasia
Brief Title: Comparison of Human Papillomavirus Integrated DNA and Messenger RNA in Cervical Neoplasia
Status: Completed | Type: Observational
Sponsor: Cathay General Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, Chih-Ming Ho, Attending physician, Cathay General Hospital
Other Study IDs: TGOG-128
Record Dates: First submitted 2009-01-04; First posted 2014-07-23 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Cervical Intraepithelial Neoplasia
Keywords: mRNA,; DNA,; integrated HPV DNA; human papillomavirus,; cervical neoplasia
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — HPV DNA and mRNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 2: Group 1: normal pap smear Group 2: cervical neoplasia

SUMMARY:
The investigators hypothesis is HPV integration could result in expression of oncogene transcripts, and not only constitutive expression but also the level of expression will be decisive for transformation and the maintenance of the malignant phenotype. Moreover, the expression and level of HPV viral transcripts not HPV DNA viral loads is correlated to the severity in cervical intraepithelial neoplasia (CIN) and cervical carcinomas (CxCa).

DETAILED DESCRIPTION:
In the investigators proposal, the investigators will examine at least 250 baseline liquid-based cytology specimens from women with normal cytology, low-grade squamous intraepithelial lesions (LSILs), high-grade squamous intraepithelial lesions (HSILs), microinvasions and invasive cervical cancers. Specimens will be tested for HPV DNA using HPV blot and type-specific PCR including type 16, 18, 52, 58, 31, 33, 39, 45, 51, 56, 59, 68, 6, and 11. Cervical specimens from women with HPV DNA types 16, 18, 52, 58, 31 and 33, which are the most prevalent oncogenic types in Taiwan, will be examined for physical status of viral DNA tested by real-time PCR and FISH, along with level of expression in mRNA.

ELIGIBILITY:
Inclusion Criteria:

* cervical neoplasia

  * HPV infection patient

Exclusion Criteria:

* no HPV infection

  * no intra-epithelial neoplasia lesion

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will examine 250 baseline liquid-based cytology specimens from women with 100 low-grade squamous intraepithelial lesions (LSILs), 100 high-grade squamous intraepithelial lesions (HSILs), 10 microinvasions and 40 invasive cervical cancers.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2007-01; Primary Completion 2009-01 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
level of mRNA expression | 12 month

SECONDARY OUTCOMES:
The integrated HPV DNA | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Ming Ho, Study Chair — Gynecologic Cancer Center, Cathay General Hospital
Locations (1):
- Cathay General Hospital, Taipei, Taiwan